CLINICAL TRIAL: NCT06274255
Title: Balikesir University, Faculty of Medicine
Brief Title: Serum Magnesium Level and Pediatric Migraine
Acronym: Migraine
Status: Not yet recruiting | Type: Observational
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Aysen Orman, Associate Prof, Mersin University
Other Study IDs: BalikesirU
Record Dates: First submitted 2024-02-05; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Migraine, Magnesium, Pediatric
Keywords: Migraine, magnesium, pediatric
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Controlle group: healthy children presenting to the pediatric neurology clinic at the same times were enrolled as the control group. The demographic characteristics (age, sex, and body mass index) of the patient group and their clinical (attack durations and frequencies, symptoms during attacks, and treatments) and laboratory (hemoglobin (Hb), hematocrit (Hct), platelet, glucose, calcium (Ca), magnesium (Mg), vitamin D, folate and ferritin levels) characteristics were recorded.
- Patients diagnosed with migraine were included as the study group: Patients diagnosed with migraine were included as the study group The demographic characteristics (age, sex, and body mass index) of the patient group and their clinical (attack durations and frequencies, symptoms during attacks, and treatments) and laboratory (hemoglobin (Hb), hematocrit (Hct), platelet, glucose, calcium (Ca), magnesium (Mg), vitamin D, folate and ferritin levels) characteristics were recorded.
  Patients and controls in whom Mg therapy was contraindicated (renal failure or nephrolithiasis), with non-migraine headaches, with substance/drug addiction (abuse), with psychiatric and/or chronic systemic diseases, and cases with histories of drug use (antidepressants, neuroleptics, tranquilizer group, antiepileptic medications (lithium and carbamazepine), using headache prophylaxis (beta blockers and calcium antagonists), and patients with deficient file data were excluded from the study.

SUMMARY:
Aim: The purpose of this study is to compare serum magnesium levels between patients with migraine and a control group and to examine the relationship between the frequency and duration of attacks in patients with migraine and mean serum magnesium levels.

Material-Method: Patients diagnosed presenting to the Balıkesir University Medical Faculty pediatric neurology clinic between 01.09.2019 and 01.04.2023 and diagnosed with migraine were enrolled retrospectively. Patients diagnosed with migraine were included as the study group and healthy children presenting to the pediatric neurology clinic in the same period as the control group. The demographic characteristics (age, sex, and body mass index) of the patient group and their clinical (attack durations and frequencies, symptoms during attacks, and treatments) and laboratory (hemoglobin, hematocrit, platelet, glucose, calcium, magnesium, vitamin D, folate and ferritin levels) characteristics were recorded.

DETAILED DESCRIPTION:
Patients diagnosed presenting to the Balıkesir University Medical Faculty pediatric neurology clinic, Türkiye, between 01.09.2019 and 01.04.2023 and diagnosed with migraine were included retrospectively. The study was approved by the institutional clinical research ethics committee (decision no. 2023/68 dated 10.05.2023).

Patients diagnosed with migraine were included as the study group and healthy children presenting to the pediatric neurology clinic at the same times were enrolled as the control group. The demographic characteristics (age, sex, and body mass index) of the patient group and their clinical (attack durations and frequencies, symptoms during attacks, and treatments) and laboratory (hemoglobin (Hb), hematocrit (Hct), platelet, glucose, calcium (Ca), magnesium (Mg), vitamin D, folate and ferritin levels) characteristics were recorded.

Patients and controls in whom Mg therapy was contraindicated (renal failure or nephrolithiasis), with non-migraine headaches, with substance/drug addiction (abuse), with psychiatric and/or chronic systemic diseases, and cases with histories of drug use (antidepressants, neuroleptics, tranquilizer group, antiepileptic medications (lithium and carbamazepine), using headache prophylaxis (beta blockers and calcium antagonists), and patients with deficient file data were excluded from the study.

Statistical analysis Descriptive characteristics (mean, number, and percentage) were determined for the study variables. Normality of distribution of numerical variables was checked. Whether continuous variables are normally distributed or not was evaluated by Kolmogorov Smirnov. Independent sample t test was used for normally distributed continuous variables. The Kruskal Wallis test was used to determine the difference between the means of three or more groups in non-normally distributed groups. Qualitative data were given as absolute reference and percentage distributions, and quantitative variables as mean and standard deviation (SD) in case of normal distribution. Categorical variables were compared using the chi-square test. Analyses were performed on Statistical Package for Social Sciences version 25 software. p values <0.05 were considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with migraine were included as the study group and healthy children presenting to the pediatric neurology clinic at the same times were enrolled as the control group.

Exclusion Criteria:

* Patients and controls in whom Mg therapy was contraindicated (renal failure or nephrolithiasis), with non-migraine headaches, with substance/drug addiction (abuse), with psychiatric and/or chronic systemic diseases, and cases with histories of drug use (antidepressants, neuroleptics, tranquilizer group, antiepileptic medications (lithium and carbamazepine), using headache prophylaxis (beta blockers and calcium antagonists), and patients with deficient file data were excluded from the study.

Ages: 72 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients diagnosed presenting to the Balıkesir University Medical Faculty pediatric neurology clinic, Türkiye, between 01.09.2019 and 01.04.2023 and diagnosed with migraine were included retrospectively. The study was approved by the institutional clinical research ethics committee (decision no. 2023/68 dated 10.05.2023).
  Patients diagnosed with migraine were included as the study group and healthy children presenting to the pediatric neurology clinic at the same times were enrolled as the control group. The demographic characteristics (age, sex, and body mass index) of the patient group and their clinical (attack durations and frequencies, symptoms during attacks, and treatments) and laboratory (hemoglobin (Hb), hematocrit (Hct), platelet, glucose, calcium (Ca), magnesium (Mg), vitamin D, folate and ferritin levels) characteristics were recorded.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-04-10 (Estimated); Study Completion 2024-05-15 (Estimated)

PRIMARY OUTCOMES:
Serum Magnesium Level and Pediatric Migraine | between 01.09.2019 and 01.04.2023
  To detect serum magnesium level in migraine attacks in children

SECONDARY OUTCOMES:
Serum Magnesium Level and Pediatric Migraine | between 01.09.2019 and 01.04.2023
  Determining serum magnesium level in children with and without migraine

CONTACTS AND LOCATIONS:
Overall Officials: Hilal Aydın, assoc. Dr., Study Director — Balikesir University
Locations (3):
- Turkey (Türkiye) (3):
  - Hilal Aydın, Balıkesir, Türkiye
  - Aysen Orman, Mersin, Türkiye
  - MersinU, Mersin, Türkiye